CLINICAL TRIAL: NCT02631811
Title: Impact on Quality of Life of an Early Management Supportive Care of Patients With Acute Leukemia in First Relapse.
Brief Title: Early Palliative Care in Patient With Acute Leukaemia
Acronym: Pablo Hemato
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL15_0305
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Leukaemia in Relapse
Keywords: acute leukaemia; supportive / palliative care
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supportive /palliative care intervention (Experimental): patients will be supported by a multidisciplinary palliative specialist team
  Interventions: Other: Supportive /palliative care intervention
- usual medical follow up (No Intervention): patients will be supported by the support care team if asked by the oncologist

INTERVENTIONS:
Other: Supportive /palliative care intervention — patients will be seen by palliative care team at least once a month until the 12th week, more if needed. The symptom and suffering will be assessed by a multidisciplinary palliative specialist team of physician, nurse and psychologist. Physical, psychological, social and existential suffering will be addressed.
  Arms: Supportive /palliative care intervention

SUMMARY:
Several studies have shown that patients with acute leukemia have many symptoms during disease These symptoms decrease the quality of life and may even appear or worsen other symptoms such as depression Several studies point to the involvement of supportive care and palliative care is delayed in these patients The aim of this study is to evaluate the impact on the quality of life of an early and standardized involvement of a support / palliative care team for patients with acute leukemia in first relapse compared to a control group .

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* acute lymphoblastic or myeloblastic leukemia at first relapse and diagnosed within 8 weeks before inclusion.
* Patients in whom a curative strategy (transplant) is not considered.
* patients older that 75 years at the diagnosis
* informed signed consent

Exclusion Criteria:

* unable to answer the questionnaire
* psychiatric disorders other than depression
* persons under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
mesure of quality of life | 12 weeks
  Quality of life measured by FACT Leu questionnaire. score of quality of life will be compared between the 2 groups

SECONDARY OUTCOMES:
measure of symptoms intensity | 12 weeks
  Symptom intensity measured by ESAS questionnaire. Score of symptoms intensity will be compared between the 2 groups
measure of depression | 12 weeks
  score of depression measured by HADS questionnaire. Score of depression will be compared between the 2 groups
measure of anxiety | 12 weeks
  score of anxiety measured by HADS questionnaire. score of anxiety will be compared between the 2 groups
measure of the quality of the end of life | up to 9 months
  Within the last month of life, several parameters will be studied to evaluate the quality of the end of life like number of admission in emergency unit.
overall survival | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier LYON SUD, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledoux M, Rhondali W, Lafumas V, Berthiller J, Teissere M, Piegay C, Couray-Targe S, Schott AM, Bruera E, Filbet M. Palliative care referral and associated outcomes among patients with cancer in the last 2 weeks of life. BMJ Support Palliat Care. 2019 Mar;9(1):e16. doi: 10.1136/bmjspcare-2014-000791. Epub 2015 Sep 23. PMID 26399699